CLINICAL TRIAL: NCT03413449
Title: A Prospective Study Frailty for Esophagectomy and Lung Resection in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1708
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Thoracic; Thoracic Neoplasm; Lung Cancer; Esophageal Cancer; Surgery--Complications; Surgery; Sarcopenia; Malnutrition; Frail Elderly Syndrome
MeSH Terms: conditions — Thoracic Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Sarcopenia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resections: Frailty model for patients undergoing esophagectomy and pneumonectomy/lobectomy for cancer
  Interventions: Diagnostic Test: Frailty model

INTERVENTIONS:
Diagnostic Test: Frailty model — 1. Grip strength
  2. 30 second chair sit stand test
  3. Psoas muscle area
  4. Six minute walk

SUMMARY:
The purpose of this study is to develop an all-encompassing frailty model using laboratory and functional studies. A frailty model will help us determine prior to surgery who will require rehabilitation and skilled nursing needs beyond discharge. This model will also help us determine who will likely be readmitted and why they will be readmitted. Understanding these things can help us prevent some of them from occurring in the future.

DETAILED DESCRIPTION:
Frailty is a widely accepted but poorly defined physical condition that has been shown to be an independent predictor of surgical morbidity and direct discharge to skilled nursing facility (SNF). Attempts have been made to study frailty in surgical patients by employing models designed for the general population. Despite the attempts of studying frailty in general surgery patients, no study has designed a model comprised of objective metrics for general thoracic surgery patients.

The purpose of this study is to better understand frailty in the context of thoracic surgery patients and to develop an objective model of this nebulous variable. It is hoped that standard, simple, functional and laboratory data can be used to construct the model with the goal being to determine the impact of frailty on outcome for patients undergoing esophagectomy, lobectomy, or pneumonectomy. If a preoperative frailty index can be developed and demonstrated to predict outcome, this scoring system may allow care teams to predict post-operative complications, ICU and hospital recidivism, and early mortality, and possibly allow for much earlier preparation for unfavorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old who are undergoing pneumonectomy, lobectomy or esophagectomy with a cancer diagnosis over a 1-year enrollment.

Exclusion Criteria:

* Patients who are unable to sign a consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with esophageal or lung cancer and are referred for surgery are included.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Morbidity | Assessed at discharge and will be reported through study completion, an average of 1 year
  Number of STS defined complications (chest tube airleak, atelectasis, pleural effusion requiring drain, pneumonia, ARDS, respiratory failure, bronchopleural fistula, PE, pneumothorax, chylothorax, ventilator > 48 hours, tracheostomy, tracheobronchial injury, ileus, anastomotic leak, GI dilation, conduit necrosis requiring surgery, delayed conduit emptying, C. diff, delirium) will be combined to report the number of morbidity events
Discharge status | Assessed at discharge and will be reported through study completion, an average of 1 year
  Discharge destination

SECONDARY OUTCOMES:
Length of stay | Assessed from date of surgery until the date of discharge and will be reported through study completion, an average of 1 year
  Time spent in the hospital during perioperative stay
30 day readmission | Assessed from date of discharge to thirty days after discharge and will be reported through study completion, an average of 1 year
  If a patient requires a readmission to the hospital within 30 days of discharge and the reasons for readmission

CONTACTS AND LOCATIONS:
Overall Officials: Sudish Murthy, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No